CLINICAL TRIAL: NCT02542202
Title: A Pilot Study of Stereotactic Body Radiotherapy (SBRT) in Oligometastatic Renal Cell Carcinoma
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Metastatic or Recurrent Kidney Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to slow enrollment
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-1542; NCI-2015-01322 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-1542 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Renal Cell Cancer; Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Stereotactic body radiation therapy (Experimental): Patients undergo stereotactic body radiation therapy on day 1 over 3 times a week for 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Undergo stereotactic body radiation therapy
  Other Names: SBRT

SUMMARY:
This pilot clinical trial studies the side effects and best dose of stereotactic body radiation therapy in treating patients with kidney cancer that has spread to other places in the body (metastatic) or has come back (recurrent). Stereotactic radiosurgery, also known as stereotactic body radiation therapy, is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or recurrent RCC (any histologic subtype)
* Patients must have between 1 to 5 new or recurrent lesions suspicious for metastatic RCC on diagnostic imaging

  * Each extracranial lesion must be =< 6 cm and amenable to SBRT or surgical excision
  * Patients must have 3 or fewer brain metastases, of size =< 4 cm

    * Brain metastases must be treated prior to enrollment in the study; the modality of treatment of brain metastases can include surgical resection, whole brain radiotherapy, stereotactic radiosurgery, or any combination of the above
  * Patients who have an intact unresected primary tumor should be considered for radical nephrectomy and primary resection prior to enrollment in the study; if the patient is not eligible for surgical resection, the primary tumor must be amenable to SBRT or request for applications (RFA); generally, this will be defined as a primary tumor < 10 cm in size or a primary lesion which can be treated to a dose of >= 8 Gy x 5 without excessive perceived risk of toxicity
* Patients must have had at least a computed tomography (CT) of the chest, abdomen, and pelvis within 4 weeks of registration in the trial; CT or magnetic resonance imaging (MRI) of the brain is only required in the presence of neurologic symptoms
* Patients must have had no radiotherapy, immunotherapy, chemotherapy or therapy with targeted agents within the last 1 month
* Patients may not have had prior bevacizumab, based on case reports of tracheoesophageal fistula in patients treated with bevacizumab and radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status =<2
* Age 18 years or older
* Life expectancy of >= 3 months
* Patients must have normal organ and marrow function within 30 days of registration, as defined below:

  * Absolute neutrophil count >= 500/mcL
  * Hemoglobin >= 8.0 g/dL
  * Platelets >= 50,000/mcL
  * Total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal if liver metastases are present
* Women of childbearing potential must have a negative pregnancy test within 14 days of registration
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior chemotherapy, immunotherapy, targeted therapy, or radiotherapy within 1 month of enrollment
* Patients who have had any prior bevacizumab, due to case reports suggesting a possible risk of severe toxicity in combination with radiotherapy
* Patients with radiographic or clinical findings of spinal cord compression or cauda equina syndrome with neurologic deficit thought to be due to malignancy
* Patients may not be receiving any systemic anti-cancer agents or other investigational agents during radiation therapy
* Patients may not have received prior radiation therapy to a site of recurrence which would require overlap of appreciable radiation dose
* Known active invasive malignancy except for renal cell carcinoma and/or non-melanoma skin cancer
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration;
  * Transmural myocardial infarction within the last 6 months prior to registration;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration;
  * Severe hepatic disease, defined as a diagnosis of Child-Pugh class B or C hepatic disease if the liver is involved with metastatic disease;
  * Human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to registration; note also that HIV testing is not required for eligibility for this protocol
* Pregnancy or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception during protocol treatment or for at least 6 months following treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Liauw, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Number of Baseline Lesions [Median (Full Range); unit: number of lesions] | 1 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiation Therapy (RT)-Related Grade >= 4 Toxicity
Description: RT-related grade >= 4 toxicity will be determined on a case-by-case basis by the study group, taking into consideration the region treated with SBRT, timing of the toxicity, and the nature of the toxicity. Rates of RT-related grade >= 4 toxicity will be recorded, time to RT-related grade >= 4 toxicity will be recorded, and freedom from RT-related grade >= 4 toxicity will be determined using the Kaplan-Meier method.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15
participants
  Skin | 0
  Nausea | 0
  Gastrointestinal | 0
  Genitourinary | 0
  Respiratory | 0
  Neurology | 0
  Total | 0

2. Secondary Outcome: Treated Lesion Control (LeC)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the start of treatment to the time of local progression at each treated lesion, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15
Participants | 1

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as defined as progression in the treated lesion, organ in which the treated lesion is present, distant failure, or death from any cause any new sites of disease on imaging or any progressive disease by RECIST criteria at initially treated sites of disease (within 80% isodose line). PFS will be estimated using descriptive statistics and the Kaplan-Meier method.
Time Frame: From start of treatment to time of progression, assessed up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of total
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15
percentage of total | 46 [20 to 68]

4. Secondary Outcome: Toxicity Profile of 5-fraction SBRT Based on Normal Tissue Dosimetric Constraints Based on the Organ Site of Involvement
Description: Toxicities of interest that occur within the 3-12 month time frame after RT start will be documented and analyzed using descriptive statistics and the Kaplan-Meier method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of total
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15
percentage of total | 85 [53 to 96]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT02542202/Prot_SAP_000.pdf